CLINICAL TRIAL: NCT02786966
Title: A Pragmatic Strategy Empowering Paramedics to Assess Low-Risk Trauma Patients With the Canadian C-Spine Rule and Selectively Transport Them Without Immobilization
Brief Title: A Pragmatic Evaluation of the Canadian C-Spine Rule by Paramedics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ontario Spor Support Unit (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CTO 0769
Record Dates: First submitted 2016-05-18; First posted 2016-06-01 (Estimated); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Neck Injuries
Keywords: Cervical spine injuries; Canadian C-spine Rule; Emergency Medical Services; Paramedic; Cervical spine fracture
MeSH Terms: conditions — Neck Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Control Phase (Other): Paramedic assessment for potential cervical spine injuries using the Canadian C-Spine Rule, but spinal immobilization using standard immobilization protocols (usual care).
  Interventions: Other: Canadian C-Spine Rule

INTERVENTIONS:
Other: Canadian C-Spine Rule — Paramedic assessment for potential cervical spine injuries using the Canadian C-Spine Rule

SUMMARY:
Each year, half a million patients with a potential neck (c-spine) injury are transported to Ontario emergency departments (ED). Less than 1% of all these patients actually have a neck bone fracture. Even less (0.5%) have a spinal cord injury or nerve damage. These injuries usually occur at the time of initial trauma and not during transport to the ED. Currently, paramedics transport all trauma victims (with or without an injury) by ambulance using a backboard, collar, and head immobilizers. Trauma victims can stay immobilized for hours until an ED bed is made available or until x-rays are completed. Importantly, long immobilization is often unnecessary, it causes patient discomfort and pain, decreases community access to paramedics, contributes to ED crowding, and is very costly.

The investigators developed the Canadian C-Spine Rule (CCR) for alert and stable trauma patients. This decision rule helps ED physicians and triage nurses to safely and selectively remove immobilization, without x-rays and missed injury.

The investigators will evaluate the possibility and benefits of allowing paramedics to use the CCR in the field in 12 new communities from across Ontario. Patients have suggested the investigators include measures of pain and discomfort from being immobilized during transport as important patient-centred outcomes. The investigators will also measure the impact on the ED, and how much money could be saved if more paramedics were allowed to use the CCR. The investigators will also assess if sex, age, language barriers, or living far from the hospital (long transport time) will affect the outcomes of the study.

DETAILED DESCRIPTION:
Paramedics in participating Ontario communities will all receive standardized training on the application of the Canadian C-Spine Rule (CCR). Once the training has been completed, paramedics will begin using the CCR to evaluate patients with potential c-spine injuries. For the first three months of the evaluation period, paramedics will use the CCR to evaluate eligible patients, but continue to use spinal immobilization for transport according to their existing protocols. After this validation period, participating services will be randomized in stepped wedge fashion in clusters of 4 services to actively use the CCR and selectively immobilize according to the CCR.

ELIGIBILITY:
Inclusion Criteria:

* Alert (Glasgow Coma Scale 15)
* Stable: Adult (16+): systolic blood pressure greater than or equal to 90 mmHg, respiratory rate 10-24 breaths/minute; Child (8-15): systolic blood pressure greater than or equal to 90 mmHg + (2 X age in years), respiratory rate 14-20 breaths/minute
* Acute blunt injury (within 48 hours of paramedic contact)

Exclusion Criteria:

* Age <8 years of age
* Penetrating trauma from stabbing or gunshot wound
* Acute paralysis (paraplegia, quadriplegia)
* Known vertebral disease (ankylosing spondylitis, rheumatoid arthritis, spinal stenosis, previous c-spine surgery)
* Referred from another hospital

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3646 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Vaillancourt, MD, MSc, Principal Investigator — Ottawa Hospital Research Insitute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vaillancourt C, Charette M, Taljaard M, Thavorn K, Hall E, McLeod B, Fergusson D, Brehaut J, Graham I, Calder L, Ramsay T, Tugwell P, Kelly P, Cheskes S, Saskin R, Plint A, Osmond M, Macarthur C, Straus S, Rochon P, Prud'homme D, Dahrouge S, Marlin S, Stiell IG. Pragmatic Strategy Empowering Paramedics to Assess Low-Risk Trauma Patients With the Canadian C-Spine Rule and Selectively Transport Them Without Immobilization: Protocol for a Stepped-Wedge Cluster Randomized Trial. JMIR Res Protoc. 2020 Jun 1;9(6):e16966. doi: 10.2196/16966. PMID 32348267

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Paramedic Services
Groups:
- Sequence 1: Usual Care Months 1-3, Canadian C-Spine Rule Months 4-9: Paramedic assessment for potential cervical spine injuries using the Canadian C-Spine Rule, but spinal immobilization using standard immobilization protocols (usual care) for months 1-3. Use of the Canadian C-Spine Rule to determine need for spinal immobilization for months 4-9.
- Sequence 2: Usual Care Months 1-6, Canadian C-Spine Rule Months 7-9: Paramedic assessment for potential cervical spine injuries using the Canadian C-Spine Rule, but spinal immobilization using standard immobilization protocols (usual care) for months 1-6. Assessment using Canadian C-Spine Rule to determine need for spinal immobilization for transport for months 7-9.
- Sequence 3: Usual Care Months 1-9: Paramedic assessment for potential cervical spine injuries using the Canadian C-Spine Rule, but spinal immobilization using standard immobilization protocols (usual care) for months 1-9.
Period: Step 1: Months 1-3
Arm/Group | Sequence 1: Usual Care Months 1-3, Canadian C-Spine Rule Months 4-9 | Sequence 2: Usual Care Months 1-6, Canadian C-Spine Rule Months 7-9 | Sequence 3: Usual Care Months 1-9
Started | 351; 4 Paramedic Services | 285; 4 Paramedic Services | 169; 3 Paramedic Services
Completed | 351; 4 Paramedic Services | 285; 4 Paramedic Services | 169; 3 Paramedic Services
Not Completed | 0; 0 Paramedic Services | 0; 0 Paramedic Services | 0; 0 Paramedic Services
Period: Step 2: Months 4-6
Arm/Group | Sequence 1: Usual Care Months 1-3, Canadian C-Spine Rule Months 4-9 | Sequence 2: Usual Care Months 1-6, Canadian C-Spine Rule Months 7-9 | Sequence 3: Usual Care Months 1-9
Started | 758; 4 Paramedic Services | 471; 4 Paramedic Services | 244; 3 Paramedic Services
Completed | 758; 4 Paramedic Services | 468; 4 Paramedic Services | 244; 3 Paramedic Services
Not Completed | 0; 0 Paramedic Services | 3; 0 Paramedic Services | 0; 0 Paramedic Services
Period: Step 3: Months 7-9
Arm/Group | Sequence 1: Usual Care Months 1-3, Canadian C-Spine Rule Months 4-9 | Sequence 2: Usual Care Months 1-6, Canadian C-Spine Rule Months 7-9 | Sequence 3: Usual Care Months 1-9
Started | 552; 4 Paramedic Services | 591; 4 Paramedic Services | 225; 3 Paramedic Services
Completed | 552; 4 Paramedic Services | 589; 4 Paramedic Services | 224; 3 Paramedic Services
Not Completed | 0; 0 Paramedic Services | 2; 0 Paramedic Services | 1; 0 Paramedic Services

BASELINE CHARACTERISTICS:
Groups:
- Control Phase (Usual Care): Paramedic assessment for potential cervical spine injuries using the Canadian C-Spine Rule, but spinal immobilization using standard immobilization protocols (usual care).
- Canadian C-Spine Rule: Assessment using Canadian C-Spine Rule to determine need for spinal immobilization for transport.
- Total: Total of all reporting groups
Arm/Group | Control Phase (Usual Care) | Canadian C-Spine Rule | Total
Number analyzed (Participants) | 1745 | 1901 | 3646
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (21.9) | 46.5 (21.9) | 47.2 (21.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 876 | 998 | 1874
  Male | 869 | 903 | 1772
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Ontario Canada
  participants
    Canada | 1745 | 1901 | 3646

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Transported With Spinal Immobilization
Time Frame: Through study completion.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Phase (Usual Care) | Canadian C-Spine Rule
Number analyzed (Participants) | 1740 | 1885
Participants | 1334 | 813
Statistical Analysis 1: Comparison: Control Phase (Usual Care) vs Canadian C-Spine Rule; Test type: Superiority; p = 0.0007, Regression, Logistic; Adjusted for age and sex; Odds Ratio (OR) = 0.4, 95% CI 2-sided [0.2 to 0.6]

2. Primary Outcome: Proportion of Patients Feeling Uncomfortable
Description: Measured on an ordinal scale from 1 to 10, with higher values indicating increasing discomfort. Values >=5 were considered to indicate discomfort.
Time Frame: At study completion
Measure: Count of Participants; unit: Participants
Arm/Group | Control Phase (Usual Care) | Canadian C-Spine Rule
Number analyzed (Participants) | 1285 | 1108
Participants | 883 | 654
Statistical Analysis 1: Comparison: Control Phase (Usual Care) vs Canadian C-Spine Rule; Test type: Superiority; p = 0.0007, Regression, Logistic; Odds Ratio (OR) = 0.61, 95% CI 2-sided [0.47 to 0.80]; Adjusted for age and sex

3. Other Pre Specified Outcome: Proportion of Patients With a Pain Score </= 5/10
Description: Measured on a 10-point ordinal scale with increasing values indicating greater pain.
Time Frame: At study completion
Measure: Count of Participants; unit: Participants
Arm/Group | Control Phase (Usual Care) | Canadian C-Spine Rule
Number analyzed (Participants) | 1423 | 1333
Participants | 866 | 736
Statistical Analysis 1: Comparison: Control Phase (Usual Care) vs Canadian C-Spine Rule; Test type: Superiority; p = 0.0093, Regression, Logistic; adjusted for age and sex; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.52 to 0.91]

4. Other Pre Specified Outcome: Time From Paramedic Arrival at Patient Side to ED Discharge or Admission to Hospital
Description: Time from paramedic arrival at patient side to ED discharge or admission to hospital
Time Frame: At time of initial injury
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Radiation Exposure
Description: radiation exposure from diagnostic imaging tests of the spine conducted at initial visit or within 30 days of the initial visit
Time Frame: 30 days from initial injury
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Number of Skin Pressure Injuries
Time Frame: through study completion (one year)
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Number of Missed Cervical Spine Injuries
Time Frame: through study completion (one year)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Paramedic Field Time (Arrival at Patient Side Until Departure for Hospital)
Description: arrival at patient side until departure for hospital
Time Frame: at time of initial injury
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Paramedic Hospital Time
Description: from arrival at emergency department to transfer of care to emergency department staff
Time Frame: through study completion (one year)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Subsequent Emergency Department Visits or Hospital Admissions
Description: within 30 days of initial visit
Time Frame: through study completion (one year)
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Subsequent Clinic or Family Physician Visits
Description: within 30 days of initial visit
Time Frame: within 30 days of initial injury
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Frequency of Cervical Spine Diagnostic Imaging
Description: at initial visit or within 30 days of initial visit
Time Frame: within 30 days of initial injury
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Cost Savings
Description: incremental cost saving per one immobilization avoided
Time Frame: through study completion (one year)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 days from time of initial paramedic assessment
Arm/Group | Control Phase (Usual Care) | Canadian C-Spine Rule
All-Cause Mortality (participants affected / at risk) | 0/1745 | 0/1898
Serious Adverse Events (participants affected / at risk) | 0/1745 | 0/1898
Other Adverse Events (participants affected / at risk) | 0/1745 | 0/1898

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT02786966/Prot_SAP_000.pdf